CLINICAL TRIAL: NCT00343187
Title: A Phase II, Randomized, Double-Blind, Parallel Design Study to Evaluate ACZONE™ (Dapsone) Gel, 5% As a Treatment For Rash Related to the Human Epidermal Growth Factor Receptor 1 (HER1)/Epidermal-Growth-Factor-Receptor (EGFR) Inhibitor Tarceva® (Erlotinib)
Brief Title: A Phase II Study of ACZONE™ (Dapsone) Gel, 5% As a Treatment For Tarceva® (Erlotinib)Related Rash
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACZ EGFR 01
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Rash; Non-small-Cell Lung Cancer
Keywords: Tarceva; Rash; EGFR-1 Rash; erlotinib; Aczone; Dapsone; Non-small Cell Lung Cancer; subjects treated with Tarceva for non-small cell lung cancer (NSCLC) who subsequently develop a rash suspected to be related to Tarceva
MeSH Terms: conditions — Exanthema; Carcinoma, Non-Small-Cell Lung | interventions — Dapsone; Gels

INTERVENTIONS:
Drug: ACZONE (dapsone) Gel, 5%
Drug: Vehicle Control

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of ACZONE in subjects treated with the HER1/EGFR inhibitor Tarceva (erlotinib) who develop a rash on the face

DETAILED DESCRIPTION:
This will be a randomized, double-blind, parallel design study in subjects treated with Tarceva for non-small cell lung cancer (NSCLC) who subsequently develop a rash suspected to be related to Tarceva. Only subjects who are not glucose-6-phosphate dehydrogenase (G6PD) deficient, and who have locally advanced or metastatic NSCLC and have failed at least 1 prior chemotherapy regimen indicated for Tarceva treatment will be included. Subjects will be screened and consented for the study within 3 days of initiating Tarceva therapy and will be instructed to contact the Investigator immediately when signs or symptoms of rash appear on the face. Subjects will be enrolled into the study only if a rash develops on the face and it has been confirmed and evaluated against eligibility criteria for the study.

Once enrolled, subjects will be randomly assigned to apply either ACZONE or placebo to the rash-affected areas of the face. Subjects will apply ACZONE / placebo treatment for 8 weeks, even if symptoms of the rash resolve completely. Specific efficacy assessments will include lesion counts, plaque area, erythema assessment, and pruritus assessment. Rash characteristics will be monitored using National Cancer Institute (NCI) Common Terminology Criteria Adverse Event (CTCAE) version 3.0 terms and severity descriptions and percentage of facial surface area (FSA) affected. Investigators will evaluate the subject's overall response to treatment according to a standardized multiple choice question. Throughout the study, photographs of the face will be taken.

Safety will be followed for 10 weeks (8 weeks of therapy + 2 weeks of follow-up) by monitoring adverse events, concomitant medications, and chemistry and hematology parameters. Plasma dapsone and N-acetyl dapsone concentrations will be measured to determine systemic exposure to the study treatment. Steady state plasma concentrations of erlotinib will also be measured before and after initiating the study treatment to determine any potential effects of ACZONE on pharmacokinetics of Tarceva.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must fulfill all of the following criteria:

1. Be male or female ≥18 years of age (inclusive).
2. Have been prescribed Tarceva as a single agent to treat locally advanced or metastatic NSCLC, after failing at least 1 prior chemotherapy regimen.
3. Present with acute signs and symptoms of rash on the face that meet the following criteria:

   1. Are suspected to be related to Tarceva,
   2. Include at least 3 inflammatory lesions, and
   3. Are less than CTCAE Grade 3 in severity.
4. Have an Eastern Co-operative Oncology Group (ECOG) performance status ≤2 and a life expectancy of at least 4 months.
5. Sign an approved informed consent form for the study.
6. Be willing to comply with the protocol.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. A skin examination reveals the presence of another skin disease and/or condition (excessive facial hair, excessive scarring, sunburn, or other disfigurement) located on the face that, in the study physician's opinion, would confound the evaluation of the rash.
2. A diagnosis of G6PD deficiency, defined as having a G6PD value below the lower limit of normal.
3. A diagnosis of anemia, defined as hemoglobin <9.5 g/dL.
4. Undergoing any current therapy for NSCLC other than Tarceva.
5. Prior treatment with Iressa, Erbitux, or any experimental HER1/EGFR inhibitor.
6. Treatment with topical antibiotics, topical steroids, and other topical treatments on the face within 14 days of Day 0 (start of ACZONE/placebo study treatment).
7. Treatment with any systemic antibiotics within 7 days of Day 0 (start of ACZONE/placebo study treatment).
8. Treatment with any systemic medication or therapy known to affect anti-inflammatory responses within 30 days prior to Day 0 (start of ACZONE/placebo study treatment). These medications include, but are not limited to, oral corticosteroids, cyclosporine, and methotrexate. Short-term treatment with non-steroidal anti-inflammatory drugs (NSAIDs) before the study for non-rash related conditions is acceptable, provided that exposure is limited to ≤7 days per course. Chronic low-dose aspirin use is also acceptable.
9. Active participation in an experimental therapy study or received experimental therapy within 30 days of Day 0 (start of ACZONE/placebo study treatment).
10. A history of hypersensitivity to dapsone, sulfamethoxazole, trimethoprim, parabens, or any component of ACZONE.
11. A poor medical risk because of other systemic diseases or active uncontrolled infections.
12. Women who: are lactating; have a positive pregnancy test at Day 0, or; if sexually active and menstruating, are not practicing an adequate method of birth control. Acceptable methods of birth control include intrauterine device (IUD); oral, dermal ("patch"), implanted or injected contraceptives; tubal ligation or hysterectomy (medical documentation required); and/or barrier methods with spermicide. A surgically sterile partner is not considered an adequate method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events; laboratory parameters; Vital signs; Pharmacokinetics

SECONDARY OUTCOMES:
Efficacy: Lesion counts; Plaque area; % of FSA affected; Erythema Score; Pruritus VAS Score; CTCAE v3.0 Grade for rash; Proportion of subjects who have rash on the face that worsens to specific category.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Garrett, MS, DDS, Study Director — QLT USA, Inc
Locations (3):
- United States (3):
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: QLT Inc. Home Page — http://www.qltinc.com